CLINICAL TRIAL: NCT04158258
Title: A STUDY TO OBSERVE PATIENTS CHARACTERISTICS, TREATMENT PATTERNS AND OUTCOMES IN PATIENTS WITH NEWLY DIAGNOSED BREAST CANCER IN LATIN AMERICA
Brief Title: A Study to Describe the Diagnosis, Anti-Cancer Treatment and Clinical Outcome in Patients With Newly Diagnosed Breast Cancer in Latin America
Status: Active, not recruiting | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Latin American Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: MO39485
Record Dates: First submitted 2019-11-05; First posted 2019-11-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Trastuzumab; Ado-Trastuzumab Emtansine; pertuzumab; atezolizumab; Capecitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (6):
- Bevacizumab: Dosing and treatment duration of any studied medicinal products collected are at the discretion of the physician in accordance with local clinical practice and local labeling.
  Interventions: Drug: Bevacizumab
- Trastuzumab: Dosing and treatment duration of any studied medicinal products collected are at the discretion of the physician in accordance with local clinical practice and local labeling.
  Interventions: Drug: Trastuzumab
- Ado-trastuzumab emtamsine: Dosing and treatment duration of any studied medicinal products collected are at the discretion of the physician in accordance with local clinical practice and local labeling.
  Interventions: Drug: Ado-trastuzumab emtamsine
- Pertuzumab: Dosing and treatment duration of any studied medicinal products collected are at the discretion of the physician in accordance with local clinical practice and local labeling.
  Interventions: Drug: Pertuzumab
- Atezolizumab: Dosing and treatment duration of any studied medicinal products collected are at the discretion of the physician in accordance with local clinical practice and local labeling.
  Interventions: Drug: Atezolizumab
- Capecitabine: Dosing and treatment duration of any studied medicinal products collected are at the discretion of the physician in accordance with local clinical practice and local labeling.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Bevacizumab — Dosing and treatment duration of any studied medicinal products collected are at the discretion of the physician in accordance with local clinical practice and local labeling.
  Other Names: Avastin
  Groups: Bevacizumab
Drug: Trastuzumab — Dosing and treatment duration of any studied medicinal products collected are at the discretion of the physician in accordance with local clinical practice and local labeling.
  Other Names: Herceptin
  Groups: Trastuzumab
Drug: Ado-trastuzumab emtamsine — Dosing and treatment duration of any studied medicinal products collected are at the discretion of the physician in accordance with local clinical practice and local labeling.
  Other Names: Kadcyla
  Groups: Ado-trastuzumab emtamsine
Drug: Pertuzumab — Dosing and treatment duration of any studied medicinal products collected are at the discretion of the physician in accordance with local clinical practice and local labeling.
  Other Names: Perjeta
  Groups: Pertuzumab
Drug: Atezolizumab — Dosing and treatment duration of any studied medicinal products collected are at the discretion of the physician in accordance with local clinical practice and local labeling.
  Other Names: Tecentriq
  Groups: Atezolizumab
Drug: Capecitabine — Dosing and treatment duration of any studied medicinal products collected are at the discretion of the physician in accordance with local clinical practice and local labeling.
  Groups: Capecitabine

SUMMARY:
A Prospective, Multicenter, Non-Interventional Study of Primary Data Collection, Designed to Describe the Diagnosis, Anti-Cancer Treatment and Clinical Outcomes in Patients with Breast Cancer in Latin America.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed newly diagnosed stage I to IV (recurrent or de novo) breast cancer no more than 12 months prior to site activation, although they can have received anti-cancer treatment during that time

Exclusion Criteria:

* Patients not receiving treatment for breast cancer with national approved drugs according to standard of care and in line with the current summary of product characteristics (SPC) /local labeling
* Patients not receiving the Roche studied medicinal product, but a biosimilar

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients will be recruited from approximately 10 countries and from a variety of healthcare sites (ex: specialty care, private practice, teaching institution, etc.)
Sampling Method: Probability Sample
Enrollment: 2907 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Different Breast Cancer Subtypes at Diagnosis in Latin America | Baseline up to 12 months

SECONDARY OUTCOMES:
Percentage of Participants with Pathological Complete Response (pCR defined ypT0/is, N0) | Baseline up to approximately 6 years
Percentage of Participants with Locoregional Recurrence (LRR) | Baseline up to approximately 6 years
Percentage of Participants with Event Free Survival (EFS) | Baseline up to approximately 6 years
Percentage of Participants with Invasive Disease-Free Survival (iDFS) | Baseline up to approximately 6 years
Percentage of Participants with Overall Survival | Baseline up to approximately 6 years
Percentage of Participants with Objective Response Rate (ORR) | Baseline up to approximately 6 years
Percentage of Participants with Anti-Cancer Treatment Modifications | Baseline up to approximately 6 years
Percentage of Participants with Breast Cancer Treatment based on Different Socio-Demographics Characteristics | Baseline up to approximately 6 years
Percentage of Participants (During Observation Period) with Pregnancy | Baseline up to approximately 6 years
Percentage of Participants (during Observation Period) with Pregnancy Outcomes | Baseline up to approximately 6 years
Percentage of Participants with Non-Serious Adverse Events of Special Interests | Baseline up to approximately 6 years
Percentage of Participants with AEs Leading to Discontinuation or Dose Modification | Baseline up to approximately 6 years
Percentage of Participants with Cardiac Safety Events | Baseline up to approximately 6 years
Percentage of Participants Adherent to Predefined Clinical Guideliens Regarding Anti-Cancer Treatment Regimens | Baseline up to approximately 6 years
Percentage of Partcipants with Access to Biomarker Testing and Diagnostic Methods | Baseline up to approximately 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (30):
- Argentina (6):
  - Instituto Alexander Fleming, Buenos Aires
  - Instituto Oncologico De Cordoba, Córdoba
  - Hospital Privado Centro Medico de Cordoba, Córdoba
  - Hospital de Morón, Morón
  - Instituto de Oncología de Rosario, Rosario
  - Sanatorio de la Mujer, Rosario
- Brazil (7):
  - Crio - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Hospital do Câncer de Londrina, Londrina, Paraná
  - Hospital Jardim Amália, Volta Redonda, Rio de Janeiro
  - Inst. de Vita, Caxias do Sul, Rio Grande do Sul
  - Centro de Pesquisa em Oncologia, Porto Alegre, Rio Grande do Sul
  - Instituto Nacional de Cancer - INCa, Rio de Janeiro
  - Instituto Brasileiro De Controle Do Câncer - IBCC, São Paulo
- Chile (3):
  - Clinica Las Condes, Santiago
  - Instituto Nacional del Cancer, Santiago
  - Hospital Dr. Hernan Henriquez Aravena, Temuco
- Colombia (4):
  - Organización Clínica Bonnadona Prevenir S.A.S, Barranquilla
  - Inst. Nacional de Cancerologia, Bogotá
  - Centro Medico Imbanaco, Cali
  - Fundacion Cardiovascular de Colombia - Instituto del Corazón, Floridablanca
- Hospital Hermanos Ameijeiras, La Habana, Cuba
- Instituto de Oncologia Dr. Heriberto Pieter, Santo Domingo, Dominican Republic
- Grupo Angeles, Guatemala City, Guatemala
- Mexico (3):
  - Instituto Nacional de Cancerologia, Mexico City, Mexico CITY (federal District)
  - Hospital Zambrano Hellion TecSalud, Monterrey, Nuevo León
  - Centro Oncologico Estatal ISSEMYM, Toluca
- Peru (3):
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
  - Clinica Internacional, Sede San Borja, Lima
  - Aliada Centro Oncologico, Lima
- Sanatorio CASMU, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: No